CLINICAL TRIAL: NCT02969226
Title: The Frequency of Screening and SBT Technique Trial: The FAST Trial, A North American Weaning Collaboration
Brief Title: The Frequency of Screening and SBT Technique Trial: The FAST Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: FAST-002
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Critically Ill
Keywords: mechanical ventilation; weaning; critically ill; spontaneous breathing trial; screening; invasive ventilation; SBT technique
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Once daily screening + PS SBTs (Active Comparator): In this arm, RTs will screen patients between approximately 06:00 - 08:00 hrs daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hrs of the scheduled screening period. Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol. RTs will conduct SBTs using only PS> 0 and =< 8 cm H2O with PEEP> 0 and =< 5 cm H2O.
  Interventions: Procedure: Once daily screening; Procedure: PS SBTs
- At least twice daily screening + PS SBTs (Experimental): In this arm patients will be screened at a minimum between approximately 06:00 - 08:00 hours and 13:00 - 15:00 hs daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hrs of the scheduled screening period. Additional screening trials in the 'at least twice daily' screening arm will be permitted at the discretion of the clinical team [RTs and physicians]. Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol. RTs will conduct SBTs using only PS>0 and =< 8 cm H2O with PEEP>0 and =< 5 cm H2O.
  Interventions: Procedure: Twice daily screening; Procedure: PS SBTs
- Once daily screening + T-piece SBTs (Active Comparator): In this arm + PS SBT' arm, RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hrs daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hrs of the scheduled screening period. Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol. RTs will conduct SBTs using only T-piece (off the ventilator).
  Interventions: Procedure: Once daily screening; Procedure: T-piece SBTs
- At least twice daily screening + T-piece SBTs (Active Comparator): In this arm, RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hours daily. If a screening period is missed inadvertently In the 'at least twice daily + PS SBT' screening arm patients will be screened at a minimum between approximately 06:00 - 08:00 hrs and 13:00 - 15:00 hrs daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hours of the scheduled screening period. Additional screening trials in the 'at least twice daily' screening arm will be permitted at the discretion of the clinical team (RTs and physicians). Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol. RTs will conduct SBTs using only T-piece (off the ventilator).
  Interventions: Procedure: Twice daily screening; Procedure: T-piece SBTs

INTERVENTIONS:
Procedure: Once daily screening — RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hours daily. To pass the 'readiness to wean screen' and undergo an SBT, specific criteria must be met.
  Arms: Once daily screening + PS SBTs; Once daily screening + T-piece SBTs
Procedure: Twice daily screening — In the 'at least twice daily' screening arm patients will be screened at a minimum between approximately 6:00-8:00 hours and 13:00-15:00 hours daily. To pass the 'readiness to wean screen' and undergo an SBT, specific criteria must be met.
  Arms: At least twice daily screening + PS SBTs; At least twice daily screening + T-piece SBTs
Procedure: PS SBTs — Patients are assigned a SBT technique. All SBTs for these patients must be conducted on PS >0 and =< 8 cm H2O with PEEP>0 and =< 5 cm H2O
  Arms: At least twice daily screening + PS SBTs; Once daily screening + PS SBTs
Procedure: T-piece SBTs — Patients are assigned a SBT technique. All SBTs for these patients must be conducted with T-piece (off the ventilator)
  Arms: At least twice daily screening + T-piece SBTs; Once daily screening + T-piece SBTs

SUMMARY:
Background: The sickest patients who are admitted to an intensive care unit (ICU) often require assistance with their breathing. When patients start to get better, they gradually do more of the breathing and the machine does less-this is called weaning. Although ventilator use saves lives, the longer it is used, the more complications can occur. Clinicians aim to wean patients from ventilators in a timely and safe manner. In most ICUs, patients are screened (looked at) once per day to see if they are ready to undergo a weaning test (using a variety of techniques) to see if the breathing tube can be removed. Screening more than once per day may allow more weaning tests to be conducted. Knowing the best way to do a weaning test is important because some methods may better determine who can have the breathing tube removed safely. At present, we don't know the best way to help our sickest patients to wean from ventilators.

Patients: Adults in North American ICUs who are on ventilators for at least 24 hours and who can take breaths on their own.

Interventions: Patients in our study will receive one type of screening and one type of weaning test at random. In the 'once daily' screening groups, clinicians will screen patients each morning. In the 'two or more times daily screening' groups, patients will be screened in the morning, afternoon, and whenever else clinicians wish to screen. When screening criteria are met, patients will undergo one of two weaning tests with low ventilator support or no support.

Outcomes: The main outcome of this study will be the time for patients to be successfully removed from the ventilator.

Relevance: For patients, this study will clarify the best way to remove them from ventilators in a timely and safe manner. For clinicians and our health care systems, this study holds promise to improve how critically ill patients are weaned from breathing machines.

DETAILED DESCRIPTION:
Goals

1. To identify the best strategy to wean patients from ventilators.
2. To fully engage patients and family members (PFM) in our trial.

Rationale: Nearly 40% of the time on invasive ventilation is spent weaning. In minimizing patients' exposure to invasive ventilation, clinicians are challenged by a trade-off between the complications associated with protracted ventilation and the risks [ventilator-associated pneumonia (VAP), mortality] of premature, failed attempts at extubation. Although randomized trials have been conducted to evaluate different screening practices and spontaneous breathing trial (SBT) techniques, most trials were small, predated daily screening, and have limited generalizability to the North American (NA) context where weaning involves respiratory therapists (RTs) and physicians.

In a systematic review of 17 trials (n=2,434), we found that screening protocols, compared to usual care, were associated with a 26% reduction in total duration of ventilation, a 70% reduction in weaning time, and an 11% reduction in ICU stay. Only 1 trial (n=385) compared twice daily screening to usual care and found that patients screened twice daily spent significantly less time on ventilators. Once daily screening is poorly aligned with the continuous care ICU environment. In our international survey, Pressure Support (PS) with positive end-expiratory pressure (PEEP) and T-piece were the most commonly used SBT techniques. Concerns exist that PS and T-piece SBTs may over and underestimate, respectively, patients' ability to breathe after extubation. Only 1 trial (n=484) has compared T-piece and PS SBTs and found no difference in outcomes. This trial was conducted in Europe, predated daily screening, and was underpowered.

Design: The investigators will conduct a factorial design trial involving 760 patients in 20 NA ICUs.

Population: The investigators will enroll critically ill adults receiving invasive ventilation for > 24 hours who can initiate or trigger breaths on commonly used weaning modes.

Comparators: Patients will be randomized to undergo a screening frequency (once vs. at least twice daily) AND an SBT technique (T-piece vs. PS ± PEEP).

Outcomes: The primary outcome will be the time to successful extubation. Secondary outcomes will include general and ventilation-specific outcomes that are important to citizens. We expect that more frequent screening, regardless of SBT technique, will reduce time to successful extubation.

This trial will identify the best strategy to reduce the time patients spend on ventilators and in ICUs, clarify best weaning practices, enhance care delivery, and launch a new paradigm of engagement into our research.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving invasive mechanical ventilation for > or = 24 hours.
2. Capable of initiating spontaneous breaths or triggering the ventilator to give a breath on ventilator modes commonly used in the ICU.
3. Fractional concentration of inspired oxygen (FiO2) < or = 70%.
4. Positive End-Expiratory pressure (PEEP) < or = 12 cm H2O.

Exclusion Criteria:

1. Brain death or expected brain death.
2. Evidence of myocardial ischemia in the 24 hour period before enrollment. Except if current trend in troponin is downward AND it has been > or = 24 hours since last troponin peak or the patient has undergone a revascularization procedure and attending physician has no concerns regarding ongoing ischemia.
3. Received continuous invasive mechanical ventilation for > or = 2 weeks.
4. Tracheostomy in situ at the time of screening.
5. Receiving a sedative infusion(s) for seizures or alcohol withdrawal.
6. Require escalating doses of sedative agents.
7. Receiving neuromuscular blockers or who have known quadriplegia, paraplegia or 4 limb weakness or paralysis preventing active mobilization.
8. Moribund (e.g., at imminent risk for death) or who have limitations of treatment.
9. Profound neurologic deficits (e.g., post cardiac or respiratory arrest, large intracranial stroke or bleed) or Glasgow Coma Scale (GCS) < or = 6.
10. Use of ventilator modes that automate SBT conduct.
11. Currently enrolled in a confounding study that includes a weaning protocol.
12. Previous enrollment in this trial.
13. Previous SBT or are already on T-piece, or CPAP alone (without PS), or PS < or equal 8 cm H2O regardless of PEEP, or other 'SBT equivalent' settings immediately before randomization.
14. Previous extubation [planned, unplanned (e.g. self, accidental)] during the same ICU admission.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Time to successful extubation | 3-4 years
  time from randomization to successful extubation

SECONDARY OUTCOMES:
ICU mortality | 3-4 years
  during index ICU admission
Hospital and 90 day mortality | 3-4 years
  during index hospital admission
Time to first passing an SBT | 3-4 years
  from randomization to SBT
Total duration of mechanical ventilation (invasive and noninvasive), | 3-4 years
  time randomization to successful extubation
ICU length of stay | 3-4 years
  reported from index ICU admission and randomization to index ICU discharge
Hospital length of stay | 3-4 years
  reported from index hospital admission and randomization to index hospital discharge
Use of NIV after extubation | 3-4 years
  Binary - yes vs no
Adverse events (e.g., self-extubation, tracheostomy, reintubation, prolonged ventilation at d14 and d21, ICU readmission) | 3-4 years
  binary - yes vs no
HRQoL (EuroQuol EQ-5D) 6 months after randomization | 6 months after randomization
  using HRQoL questionnaire
Functional status 6 months after randomization using either the IES-R, Lawton ADL scale, or the FIM | 6 months after randomization
  using Functional status questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Karen Burns, MD, FRCPC, Principal Investigator — St. Michael's Hospital (Toronto, Canada)
Locations (16):
- United States (5):
  - Longbeach Memorial Hospital, Long Beach, California
  - Keck Hospital of USC, Los Angeles, California
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Temple University Hospital, Philadelphia, Pennsylvania
- Canada (11):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital Cancer Centre, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Niagara Health - St. Catharines, Niagara, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Universite de Sherbooke, Sherbrooke, Quebec
  - Ciusss McQ, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burns KEA, Wong J, Rizvi L, Lafreniere-Roula M, Thorpe K, Devlin JW, Cook DJ, Seely A, Dodek PM, Tanios M, Piraino T, Gouskos A, Kiedrowski KC, Kay P, Mitchell S, Merner GW, Mayette M, D'Aragon F, Lamontagne F, Rochwerg B, Turgeon A, Sia YT, Charbonney E, Aslanian P, Criner GJ, Hyzy RC, Beitler JR, Kassis EB, Kutsogiannis DJ, Meade MO, Liebler J, Iyer-Kumar S, Tsang J, Cirone R, Shanholtz C, Hill NS; Canadian Critical Care Trials Group. Frequency of Screening and Spontaneous Breathing Trial Techniques: A Randomized Clinical Trial. JAMA. 2024 Dec 3;332(21):1808-1821. doi: 10.1001/jama.2024.20631. PMID 39382222